CLINICAL TRIAL: NCT04891120
Title: Treadmill Stress Test With and Without Mask: Comparison of Exercise Capacity and Perception
Brief Title: Treadmill Stress Test With and Without Mask
Acronym: TREADMASK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2021-4210
Record Dates: First submitted 2021-05-05; First posted 2021-05-18 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Healthy
Keywords: Treadmill; Bruce; COVID-19; Mask; Healthy; Adults; METS; Metabolic equivalent; Borg; Exercise; Stress test
MeSH Terms: conditions — Brucellosis; COVID-19; Motor Activity | interventions — Exercise Test

STUDY DESIGN:
Masking Description: The statistician will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- With, then without a mask (Experimental): Participants will first perform a treadmill test with a mask and 48 hours or more later will perform another similar treadmill test without a mask.
  Interventions: Diagnostic Test: Treadmill test (Bruce protocol)
- Without, then with a mask (Experimental): Participants will first perform a treadmill test without a mask and 48 hours or more later will perform another similar treadmill test with a mask.
  Interventions: Diagnostic Test: Treadmill test (Bruce protocol)

INTERVENTIONS:
Diagnostic Test: Treadmill test (Bruce protocol) — Treadmill test performed with and without a mask.

SUMMARY:
The purpose of this study is to assess if wearing a surgical mask affects the results of a standard treadmill test.

DETAILED DESCRIPTION:
The persons interested to participate will be informed of the implication and potential risks associated with the study. The participants that accept and meet the eligibility criteria will give written consent and be randomized into two groups. One group will first perform a treadmill test with a surgical mask and then repeat the test without a mask. The second group will do the first treadmill test without a mask and the second one with a surgical mask.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18-65 years old)
* Healthy
* Vaccinated against COVID-19

Exclusion Criteria:

* Any cardiac or respiratory condition
* Walking difficulty
* Waiting for a stress test for a medical reason
* Abnormal resting ECG
* Inability to wear a mask
* Inability to understand or follow the instructions
* Medical contraindication to performing a treadmill stress test

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2021-05-11 (Actual); Primary Completion 2021-06-16 (Actual); Study Completion 2021-06-16 (Actual)

PRIMARY OUTCOMES:
Change in Metabolic Equivalents With vs Without a Mask | Through study completion, an average of 1 week
  The maximal metabolic equivalents achieved will be calculated for each treadmill test performed.

SECONDARY OUTCOMES:
Change in Borg's Category-Ratio Scale for Rating of Perceived Exertion With vs Without a Mask | Through study completion, an average of 1 week
  The Borg Scale is a self-reporting instrument assessing intensity of perceived exertion on a 0 to 10 scale, 0 being rest and 10 maximal effort.

OTHER OUTCOMES:
Change in Exercise Duration With vs Without a Mask | Through study completion, an average of 1 week
Change in Heart Rate During Exercise With vs Without a Mask | Through study completion, an average of 1 week
Change in Blood Pressure During Exercise With vs Without a Mask | Through study completion, an average of 1 week
Change in Oxygen Saturation During Exercise With vs Without a Mask | Through study completion, an average of 1 week
Change in Duration of Exercise Before Reaching 85% of Predicted Maximal Heart Rate With vs Without a Mask | Through study completion, an average of 1 week
Change in Calculated Maximal Oxygen Consumption During Exercise With vs Without a Mask | Through study completion, an average of 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Warner Mampuya, MD, PhD, Principal Investigator — Université de Sherbrooke
Locations (1):
- Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlies results in a publication will be available in the supplementary appendix of the publication or on request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will be available at the time of the publication and for the 2 following years.